CLINICAL TRIAL: NCT02181855
Title: Effect of Full-thickness Gastroplication With the GERD-X System on Atypical Gastro-esophageal-reflux-symptoms.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: atyGERD-X
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Atypical Gastroesophageal Reflux Symptoms; Objectified Gastroesophageal Reflux Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atypical GERD syptoms treated with GERD-X (Other): Patients treated by means of full-thickness gastroplication
  Interventions: Procedure: Full-thickness gastroplication (GERD-X)

INTERVENTIONS:
Procedure: Full-thickness gastroplication (GERD-X) — Endoscopic full-thickness gastroplication wit the GERD-X device

SUMMARY:
Patients with atypical symptoms of objectified gastroesophageal reflux disease will be treated by full-thickness gastroplication and the effect of this intervention will be measured by questionnaires and clinical diagnostics (for example pH/MII).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 years and 80 years
* symptomatic, objectified reflux disease (atypical symptoms - Montreal-classification)

Exclusion Criteria:

* Rejection of study-participation,
* Pregnancy
* negative pH-metry / impedance monitoring (non-objectified reflux)
* hiatal hernia bigger than 2 cm or gastroesophageal junction > Hill IV classification
* different potential reasons for atypical symptoms like heterotopic gastric mukosa in the cervikal esophagus
* Achalasia, esophageal spasm
* Presence of contraindications for the interventions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reflux Symptom index | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Monther Bajbouj, PD Dr. med., Principal Investigator — Klinikum rechts der Isar, II. Med; Simon Nennstiel, Dr. med., Principal Investigator — Klinikum rechts der Isar, II. Med
Locations (4):
- Krankenhaus der Barmherzigen Schwestern Linz, Klinik für Allgemein- und Viszeralchirurgie, Linz, Austria
- Germany (3):
  - Klinikum rechts der Isar der Technischen Universität München, II. Med. Klinik und Poliklinik, München, Bavaria
  - Klinikum rechts der Isar der Technischen Universität München, Klinik und Poliklinik für Chirurgie, München, Bavaria
  - Klinikum Ludwigsburg, Klinik für Innere Medizin, Gastroenterologie, Hämato-Onkologie, Diabetologie und Infektiologie, Ludwigsburg